CLINICAL TRIAL: NCT06156189
Title: Prevalence of Enteral Nutrition Interruption in an Oncology Intensive Care Unit. A Prospective Observational Study
Brief Title: Prevalence of Enteral Nutrition Interruption in an Oncology Intensive Care Unit.
Status: Completed | Type: Observational
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Principal Investigator, Muhammad Rehan Akram, Consultant Pulmonary Physician, King Faisal Specialist Hospital & Research Center
Other Study IDs: REC-2022- 0005
Record Dates: First submitted 2023-11-26; First posted 2023-12-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness | interventions — Enteral Nutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Critically ill patients: All adult patients ventilated and intubated. These patients should also have enteral nutritional supplement initiated.
  Interventions: Dietary Supplement: Enteral Feeding

INTERVENTIONS:
Dietary Supplement: Enteral Feeding — Feeding via Nasogastric tube in intubated and ventilated patients

SUMMARY:
This is a single-center retrospective observational study. The study aimed to look at the enteral feed interruptions in patients who were intubated and ventilated in an oncology intensive care unit. We collected data of the first 60 interruptions in the adult Oncology ICU from 12/12/2022 to 15/10/2023. We only included intubated and ventilated adult patients more than 18 years of age who had nasogastric tube feeding commenced. The data was collected from the electronic patient records. Data collected included demographics, total interruption time per episode of interruption, the reason for the delay, whether the delay could have been avoided, total calories lost, and percentage of calories lost.

DETAILED DESCRIPTION:
Introduction Intensive Care Unit (ICU) patients are often intubated and ventilated. These patients cannot feed themselves orally, so enteral or parenteral nutrition becomes important. Various studies have suggested that meeting their nutritional demand is associated with their short and long-term outcomes. There is also ample evidence that in general ICU's, patients often do not meet their nutritional demands. (1,2) The ICU may often differ in the nature of the patients catered for and also may have very different systems of delivering healthcare provisions. This could have an impact on the patient care provided.

There are several studies suggesting that EN interruptions happen frequently in the ICU. (3,4,5) It is estimated that the EN interruption occurs in more than 85% of the patients for an average of 8-20% of the infusion time. Out of this, it is thought that 23% are avoidable in planned procedures and 65% on all occasions. (6) There is very little data on the duration of the interruptions and those associated with diagnostic procedures.

In this single-centre study, we aim to understand the prevalence of instances of missed feeding within an oncology-focused ICU in intubated patients. We looked at the reason for the delay and estimated the calorie deficit, the duration of the delay and the proportion of patients who met at least 60% of the calorie requirement. This is an important step in developing a feeding protocol to minimize such instances.

Methods This study included all intubated patients admitted to the Intensive Care Unit at the King Faisal Specialist Hospital and Research Centre from December 2022 to November 2023. The inclusion criteria were defined as adult patients above the age of 18 who were intubated and ventilated and started on enteral feeding via nasogastric tube. All patients who were not intubated and under 18 years of age were excluded.

Data will be collected from the electronic patient records. The data collected will be demographics, diagnosis, time the feed was started and stopped, delay in restarting the feed, estimated daily calorie requirement, and calorie deficit. The daily calorie requirement will be estimated using the quick calorie method using kilocalories per kilogram Table1. To estimate the actual calorie intake of the patient, the enteral feeding flowsheet of each patient was monitored, and the total intake will be calculated (mL/hr) for the whole day and based on the type of feed (High calorie, standard etc) it will be multiplied to the total intake to get the actual calorie intake.

Energy requirements Based on Kilocalories per kilogram of body weight condition Energy requirement (kcal/kg) Normal 25-30 (kcal/kg) Obese, critically ill, (BMI>30) 11-14 (actual body weight) or 22-25 (ideal body weight) Mild stress 30-35 (kcal/kg) Moderate to severe 35-45 (kcal/kg)

Table1. The formula used for estimating calorie requirement. The calorie deficit was calculated from this. The percentage of lost calories will be tabulated, and the number of instances where patients received >60% or <60% of the daily requirement will be computed.

The local Research Ethics Committee approved the study. As the study was a non-interventional observational study, a consent waiver was requested and was approved by the ethics committee.

Statistical analysis Demographics will be analyzed for the frequency of distribution. The incidence of feed interruption will be calculated and expressed as median, mean and percentage. The proportion of lost calories and calorie deficit will be calculated in numbers and percentages. The commonest reason for delay, avoidable and unavoidable reasons for feed interruption and the proportion of patients who missed more than 60% of the estimated daily requirement will be estimated using frequencies. Spearmen's correlation rank test will be used to examine the relation between the delay in restarting feed and the lost calories.

ELIGIBILITY:
Inclusion Criteria:

- Adult patients above the age of 18 who were intubated and ventilated and started on enteral feeding via nasogastric tube

Exclusion Criteria:

* Patients less than the age of 18
* Patients not intubated and ventilated
* Patients not critically ill

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: -All adult patients who were intubated and ventilated in an adult oncology ICU
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-12-12 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Incidence of number of enteral feed interruptions | December 2022 to October 2023
  Enteral feeding interruptions

SECONDARY OUTCOMES:
Calorie deficit | December 2022 to October 2023
  Estimated daily calorie required was calculated and actual calorie received by the patient was calculated and calorie deficit was calculated from this.
Reasons Delay in restarting Enteral feeding | December 2022 to October 2023
  Reasons for stopping and restarting feed was recorded
Delay in feeding in hours | December 2022 to October 2023
  Delay in restarting the feed in hours were calculated
Avoidable and unavoidable delays | December 2022 to October 2023
  If the delays were due to factors that could be modified or not modifiable were recorded

CONTACTS AND LOCATIONS:
Locations (1):
- King Faisal Specialist Hospital and Research Centre, Al Madīnah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
As of now there is no ethical approval and reason to share individual patient details. However, the team will be able to share anonymized dataset if deemed necessary

REFERENCES:
- [Result] Nurkkala JP, Kaakinen TI, Vakkala MA, Ala-Kokko TI, Liisanantti JH. Nutrition deficit during intensive care stay: incidence, predisposing factors and outcomes. Minerva Anestesiol. 2020 May;86(5):527-536. doi: 10.23736/S0375-9393.20.14068-9. Epub 2020 Jan 28. PMID 32000472
- [Result] Uozumi M, Sanui M, Komuro T, Iizuka Y, Kamio T, Koyama H, Mouri H, Masuyama T, Ono K, Lefor AK. Interruption of enteral nutrition in the intensive care unit: a single-center survey. J Intensive Care. 2017 Aug 4;5:52. doi: 10.1186/s40560-017-0245-9. eCollection 2017. PMID 28794882
- [Result] McClave SA, Sexton LK, Spain DA, Adams JL, Owens NA, Sullins MB, Blandford BS, Snider HL. Enteral tube feeding in the intensive care unit: factors impeding adequate delivery. Crit Care Med. 1999 Jul;27(7):1252-6. doi: 10.1097/00003246-199907000-00003. PMID 10446815
- [Result] Passier RH, Davies AR, Ridley E, McClure J, Murphy D, Scheinkestel CD. Periprocedural cessation of nutrition in the intensive care unit: opportunities for improvement. Intensive Care Med. 2013 Jul;39(7):1221-6. doi: 10.1007/s00134-013-2934-8. Epub 2013 May 1. PMID 23636828